CLINICAL TRIAL: NCT04495322
Title: A Phase 1, Single-center, Randomized, Double-blind, Placebo-controlled, Single-dose Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics Profiles of TG-1000 in Healthy Volunteers, and to Evaluate the Food Effect on Pharmacokinetics of Single Oral Dose of TG-1000 in Healthy Volunteers.
Brief Title: To Evaluate the Safety, Tolerability, and Pharmacokinetics Profiles of TG-1000 in Healthy Volunteers, and the Food Effect on Pharmacokinetics of Single Oral Dose of TG-1000 in Healthy Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TaiGen Biotechnology Co., Ltd. (Industry)
Collaborators: R&G Pharma Studies Co.,Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: TG-1000-C-01
Record Dates: First submitted 2020-07-22; First posted 2020-07-31 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Healthy Chinese Volunteers

STUDY DESIGN:
Intervention Model Description: single-center, randomized, double-blind, placebo-controlled, single-dose
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- 10 mg TG-1000 (Experimental): Eligible subjects will receive single oral dose of study drug (2 x 5-mg TG-1000 capsules)on Day 1 under fasted condition.
  Interventions: Drug: TG-1000
- 20 mg TG-1000 or Placebo (Experimental): Eligible subjects will receive single oral dose of study drug (20 mg TG-1000 capsule or Placebo capsule) on Day 1 under fasted condition.
  Interventions: Drug: TG-1000; Drug: Placebo
- 40 mg TG-1000 or Placebo (Experimental): Eligible subjects will receive single oral dose of study drug (2 x 20 mg TG-1000 capsules or Placebo capsules) on Day 1 under fasted condition.
  Interventions: Drug: TG-1000; Drug: Placebo
- 80 mg TG-1000 or Placebo (Experimental): Eligible subjects will receive single oral dose of study drug (4 x 20 mg TG-1000 capsules or Placebo capsules) on Day 1 under fasted condition.
  Interventions: Drug: TG-1000; Drug: Placebo
- 120 mg TG-1000 or Placebo (Experimental): Eligible subjects will receive single oral dose of study drug (6 x 20 mg TG-1000 capsules or Placebo capsules) on Day 1 under fasted condition.
  Interventions: Drug: TG-1000; Drug: Placebo
- 160 mg TG-1000 or Placebo (Experimental): Eligible subjects will receive single oral dose of study drug (8 x 20 mg TG-1000 capsules or Placebo capsules) on Day 1 under fasted condition.
  Interventions: Drug: TG-1000; Drug: Placebo
- X mg TG-1000 (fasted)+wash-out+X mg TG-1000 (fed) (Experimental): Based on the preliminary results, one optimal dose (X mg) of TG-1000 will be selected. Subject will receive a single oral dose of TG-1000 under fasted condition. After washout period, subject will receive a single oral dose of TG-1000 under fed condition.
  Interventions: Drug: TG-1000
- X mg TG-1000 (fed)+wash-out+X mg TG-1000 (fasted) (Experimental): Based on the preliminary results, one optimal dose (X mg) of TG-1000 will be selected. Subject will receive a single oral dose of TG-1000 under fed condition. After washout period, subject will receive a single oral dose of TG-1000 under fasted condition.
  Interventions: Drug: TG-1000

INTERVENTIONS:
Drug: TG-1000 — Subjects will receive one single oral dose of TG-1000 on day 1 following protocol requirements.
Drug: Placebo — Subjects will receive one single oral dose of placebo on day 1 following protocol requirements.
  Arms: 120 mg TG-1000 or Placebo; 160 mg TG-1000 or Placebo; 20 mg TG-1000 or Placebo; 40 mg TG-1000 or Placebo; 80 mg TG-1000 or Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics profiles of TG-1000 in healthy volunteers, and to evaluate the food effect on pharmacokinetics of single oral dose of TG-1000 in healthy volunteers.

DETAILED DESCRIPTION:
This is a phase 1, single-center, randomized, double-blind, placebo-controlled, single-dose escalation study to evaluate the safety, tolerability, and pharmacokinetics profiles of TG-1000 in healthy volunteers, and to evaluate the food effect on pharmacokinetics of single oral dose of TG-1000 in healthy volunteers. The study will be divided into two parts.

Part A is designed as randomized, double-blind, placebo-controlled, sequential, single ascending oral dose to evaluate the safety, tolerability, and PK profiles of TG-1000 in healthy volunteers.

Part B is designed as randomized, open-label, two treatment (fasted vs. fed), two-period, two-sequence crossover to compare the effects of food on the Pharmacokinetic (PK) of single oral dose of TG-1000 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to provide written informed consent.
2. Age 18 (or legal adult age) to 45 years.
3. Body mass index (BMI) in the range of ≥19.0 to ≤ 24.0 kg/m2 and body weight ≥ 50 kg for male and ≥ 45 kg for female at Screening.
4. Subjects have good communication with Investigator and agree to follow the study requirement to complete study.

Exclusion Criteria:

1. Clinically significant abnormality in 12-lead ECG, chest X-ray, abdominal ultrasounds, physical examination, vital signs or laboratory values at Screening or Day-1.
2. Positive breath alcohol or urine drug tests at Day-1.
3. Positive test results for Immunoglobulin M anti-HAV antibody, HBsAg, anti-HCV antibody, HIV or syphilis at Screening.
4. Female subjects with positive pregnancy test results at Screening or Day-1.
5. Male subjects are unwilling to use effective contraception and refrain from sperm donation from Screening until 3 months after the study drug administration.
6. Current or prior history of any of the following:

   1. Significant cardiac disease, diabetes, liver, kidney disease, psychiatric diseases or drug abuse or diseases that will affect immunity.
   2. Difficulty in swallow or gastrointestinal disorder that could interfere with the absorption of the study drug
   3. Difficulty in blood sampling or venipuncture
   4. Drug allergy or hypersensitivity
   5. Blood donation ≥ 400 mL within 3 months before and after study.
   6. Alcoholics or frequent drinkers prior to Screening.
   7. Frequent smokers prior to Screening.
7. Use of any prohibited medications or surgeries prior to study drug administration:

   a. Received any other investigational agents or devices, liver enzyme inducer or inhibitors, medications including prescriptions, non-prescriptions or herbal remedies, dietary supplements or surgeries.
8. Unwilling to abstain from alcohol, tobacco, nicotine containing products, caffeine- or xanthine-containing beverages from Screening until discharge from the phase I unit.
9. Subjects may not be qualified for the study judged by the Investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2020-07-17 (Actual); Primary Completion 2020-11-26 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Number of subjects of treatment-emergent adverse events | 8 days
  Any significant findings after dosing will be considered as adverse events.
Number of subjects of Significant Abnormal Vital Signs Findings | 8 days
  The systolic and diastolic blood pressure (mmHg), pulse/heart rate (beats/min), respiratory rate (breaths/min), and body temperature (oC) will be measured.
Number of subjects With Significant Abnormal Physical Examination Findings | 8 days.
  A full general physical examination of the major body systems (General Appearance; Dermatological including skin and nails; Head and Neck; Chest region including Heart and Lung; Abdominal region including Gastrointestinal and Gastroenterology; Back region; Extremities; Psychiatric or Neurological; Lymph nodes; Other) will be performed by investigator.
Number of subjects With Significant Abnormal 12-lead Electrocardiography (ECG) Findings | 8 days
  12-lead ECG will be performed after a rest in a supine position. The following ECG parameters will be listed: heart rate, the time between QRS complexes (RR Interval) (ms), the beginning of the P wave to the first deflection of the QRS complex (PR Interval) (ms), first deflection of QRS complex to end of QRS complex at isoelectric line (QRS duration) (ms), first deflection of QRS complex to end of T wave at isoelectric line (QT interval) (ms), Corrected QT interval by Bazett (QTcB) (ms), and Corrected QT interval by - Fridericia (QTcF) (ms).
Number of subjects With Significant Abnormal Holter Electrocardiography (ECG) Findings | 12 hr pre-dose until 24 hr post-dose
  Holter ECG will be monitor continue from 12 hr pre-dose until 24 hr post-dose. The Investigator will determine whether the results of the Holter monitoring are normal or abnormal.
Number of Participants With Significant Abnormal Laboratory Values | 8 days
  Chemistry, Hematology, Coagulation, Urinalysis, Human Immunodeficiency Virus (HIV) test, Hepatitis A virus(HAV) test, Hepatitis B virus (HBV) test, Hepatitis C virus (HCV) test, syphilis, serum pregnancy tests and Breath Alcohol Test
Peak Plasma Concentration (Cmax) | 15 days
  Blood sample will be collected to evaluate PK profile and food effect of TG-1000.
time to Cmax (Tmax) | 15 days
  Blood sample will be collected to evaluate PK profile of TG-1000.
area under the curve from time zero to the time (AUC0-t) | 15 days
  Blood sample will be collected to evaluate PK profile and food effect of TG-1000.
area under the concentration-time curve from time zero to the last quantifiable concentration (AUC0-last) | 15 days
  Blood sample will be collected to evaluate PK profile of TG-1000.
area under the concentration-time curve from time zero to infinity (AUC0-inf) | 15 days
  Blood sample will be collected to evaluate PK profile and food Effect of TG-1000.
terminal elimination half-life (T1/2, z) | 15 days
  Blood sample will be collected to evaluate PK profile of TG-1000.
apparent total body clearance (CL/F) | 15 days
  Blood sample will be collected to evaluate PK profile of TG-1000.
apparent total volume distribution (V/F) | 15 days
  Blood sample will be collected to evaluate PK profile of TG-1000.
plasma concentration 24 h after dosing (C24) | 15 days
  Blood sample will be collected to evaluate PK profile of TG-1000.
urinary excretion ratio relative to dose from time zero to the time (Feu0-t) | 15 days
  Urine sample will be collected to evaluate PK profile of TG-1000.

CONTACTS AND LOCATIONS:
Overall Officials: Pingsheng Xu, Principal Investigator — Xiangya Hospital of Central South University
Locations (1):
- Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No